CLINICAL TRIAL: NCT06805409
Title: Evaluation of Venous Congestion Using Doppler and Venous Excess Ultrasound Score (VExUS) During Acute Respiratory Distress Syndrome and Its Association with Acute Kidney Injury
Brief Title: VExUS in Ards Patients and Association with AKI
Acronym: VEXAKI
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240897
Record Dates: First submitted 2024-11-05; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS)
Keywords: Acute respiratory distress syndrome; acute kidney injury; Venous Congestion
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Acute Kidney Injury; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A single-center prospective observational study will be conducted with the aim of determining the prevalence of venous congestion during ARDS using venous Doppler and the VExUS score.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is common in patients with acute respiratory distress syndrome (ARDS) and is associated with higher mortality rates. Among the mechanisms underlying this AKI, venous congestion seems to be significant. However, methods for assessing congestion are limited and may be unreliable. The use of venous Doppler (inferior vena cava, suprahepatic veins, portal vein, and intrarenal veins) for grading the severity of congestion using the Venous Excess Ultrasound Score (VExUS) could potentially enable the earlier identification of ARDS patients with congestion.

A prospective observational monocenter study will be conducted with the objective to determine the prevalence of venous congestion during ARDS using venous Doppler and the VExUS score.

The primary outcome measure will be the proportion of patients with a VExUS score ≥ 1 within 48 hours following the initiation of invasive mechanical ventilation. The secondary objective is to evaluate the association of different VExUS grades with the occurrence of the composite endpoint of major kidney events at Day 30 (MAKE-30), defined as the occurrence of death, dependence on dialysis, or persistent elevation of creatinine ≥ 200% of baseline creatinine.

The study involves adult patients admitted to the intensive care unit with moderate to severe ARDS requiring mechanical ventilation for less than 48 hours and requiring hemodynamic support with catecholamines. Within 48 hours of initiating invasive mechanical ventilation, concurrently with the cardiac ultrasound, the multi-site venous Doppler will be performed. Demographical, clinical, and biological data will be prospectively collected. The multi-site venous Doppler will be repeated on Day 7 of mechanical ventilation initiation or during catecholamine weaning, depending on which event occurs first. Patients will be followed for the entire duration of their intensive care unit stay. For patients discharged alive from the intensive care unit, follow-up will continue until 3 months after discharge to assess the occurrence of chronic kidney disease following the initial hospitalization.

No other investigations are mandated by the protocol besides performing the multi-site venous Doppler.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Moderate to severe ARDS according to the Berlin definition
* Requiring catecholamine support
* Undergoing invasive mechanical ventilation for less than 48 hours

Exclusion Criteria:

* Patients presenting with acute kidney injury KDIGO III requiring renal replacement therapy before the initial ultrasound evaluation
* Requirement for veno-venous or veno-arterial ECMO circulatory support before inclusion
* Patients with end-stage chronic kidney disease, on dialysis, and/or kidney transplant recipients
* History of Child C cirrhosis and/or liver transplantation and/or portal hypertension
* History of portal thrombosis
* Known history of pulmonary hypertension
* Pregnant women
* Patients under legal protection
* Patients who have expressed opposition to participating in the research

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study concerns adult patients hospitalized in intensive care for moderate to severe ARDS according to the Berlin definition, and requiring hemodynamic support with catecholamineEKG
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2027-12-09 (Estimated); Study Completion 2027-12-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of VExUS score ≥ 1 within 48 hours of invasive mechanical ventilation. | 48 hours, 7 days after mechanical ventilation
  Quantification of the VExUS score from the measurement of the inferior vena cava size, an assessment of suprahepatic venous flow, portal venous flow and intra-renal venous.

SECONDARY OUTCOMES:
Occurrence of the composite endpoint of major kidney events at Day 30 (MAKE-30). | 30 days
  defined as death, dependence on dialysis, or persistence of a creatinine elevation ≥ 200% of baseline creatinine.

CONTACTS AND LOCATIONS:
Locations (1):
- Armand MEKONTSO DESSAP, Créteil, Val de Marne, France